CLINICAL TRIAL: NCT04546048
Title: The Early Strength Training Exercise Therapy in Liver Recipients: Protocol for an Observational Feasibility Trial
Brief Title: The Early Strength Training Program in Post-transplant Liver Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Hospital Groups (Other)
Responsible Party: Principal Investigator, Tuba Ergene, MSc, Memorial Hospital Groups
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015970102
Record Dates: First submitted 2020-09-06; First posted 2020-09-11 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: End Stage Liver DIsease; Chronic Liver Failure; Liver Transplant Disorder; Muscle Loss; Muscle Weakness; Sarcopenia; Fatigue; Quality of Life
Keywords: muscle strength; liver transplantation; resistance training; functional status
MeSH Terms: conditions — End Stage Liver Disease; Muscular Atrophy; Muscle Weakness; Sarcopenia; Fatigue | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (EG) (Experimental): The exercise group (EG) were received an 8-week resistance training program in addition to standard post-transplant physiotherapy follow-up.
  Interventions: Behavioral: Strength Exercise Training
- Control Group (CG) (No Intervention): The control group (CG) were received only standard physiotherapy program.
  The usual post-transplant care consisting of preoperative patient education, respiratory physiotherapy program, active/active assistive exercises of cervical, upper and lower extremities, and early mobilization.
  Patients were instructed about the postoperative physiotherapy process including all details within the preoperative education. Respiratory physiotherapy consisted of positioning, lung expansion exercises and bronchial hygiene techniques.
  They were allowed to pursue their normal daily activities and mobilized as early as possible when clinically stable.

INTERVENTIONS:
Behavioral: Strength Exercise Training — The 8-week exercise-training program consisted of two 30-min sessions a day for 5 days/week and conducted by elastic exercise bands in 2-3 sets, 6-10 repetitions, with 1-2 min rest between sets (M. Deltoideus and M. Quadriceps are trained as major muscle groups). The 8-repetition maximum(8RM) is used to determine training loads with the rated perceived exertion(RPE) lower than 5-7 on the Modified Borg scale(MBS). The program consisted functional exercises by half squat to squat and sit-to-stand chair exercises. Exercise sessions were supervised twice daily during the 1st week, the 2nd week training included one supervised and one unsupervised daily sessions. The remaining 6-week training program conducted at home individually after discharge. Patients instructed for the ongoing 8-week training program and a patient-specific schedule delivered to subjects. Phone calls are provided weekly and training load is assessed while generating 4th week evaluations.
  Other Names: Resistance Training
  Arms: Exercise group (EG)

SUMMARY:
Liver transplantation (LT) is a current life-saving procedure performed as an open-abdominal surgery for patients with end-stage liver diseases (ESLD). However, a high risk of post-surgical complications is relevant to major intra-abdominal interventions. In managing post-LT recovery, it is important to consider the extending pre-transplant physical status of ESLD patients concerning an impaired exercise capacity, a prolonged period of deconditioning, fatigue and muscle weakness, which leads to global motor impairment and decreased functional capacity.

Sarcopenia and physical deconditioning are known as the hallmark features of ESLD. The quality and the quantity of skeletal muscle mass have been closely correlated with post-transplantation mortality in individuals undergoing LT. In addition to chronic deconditioning or myopathy related to chronic liver failure, post-transplant immunosuppressive medication contributes to increased risk for age-related decline in muscular strength and physical ability. It reportedly persists impaired physical function including reduced muscle strength, which have been consistently associated with impaired quality of life after a liver transplant.

Exercise interventions in solid-organ recipients provide improvements in physical function including skeletal muscle strength. The literature has defined many types of exercise-based interventions including aerobic and resistive training or physical activity counselling in improving physical performance tasks, muscle strength and physical domain of quality of life in postoperative liver transplanted adults. Although there are studies in improving muscle performance and functional status, no study conducted in the post-transplant early period and an optimal exercise regimen for post-liver recipients. In the present study, it will be provided a framework for a possible change in practice aiming to improve muscle strength and functionality in liver recipients through a strength training exercise intervention at the early post-transplant period. The purposes of this trial were: 1) to evaluate the feasibility and safety of a strength exercise training program on functional mobility and quality of life of liver transplanted individuals and 2) to initiate physiotherapy protocols in this population. A key component of this approach was that it was individualized, providing one-to-one therapy with tailored progression specific to a person's individual mobility goals.

ELIGIBILITY:
Inclusion Criteria:

* Liver recipients were eligible to participate if they were 1) over 18 years old, 2) completed the pre-operative evaluation procedure, 3) post-op hemodynamically stabled and had spontaneous breathing, 4) able to read, write and understand Turkish language.

Exclusion Criteria:

* Study exclusion criteria were having unstable cardiovascular disease, a primary lung pathology requiring regular bronchodilator treatment, neuromusculoskeletal complication and/or limitation which requiring the use of assistive device, being a multi-organ transplant recipient and difficulty in following verbal orders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-08-24 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | baseline (pre-operative), 4th and 8th post-operative week
  The measurement of the maximal inspiratory and expiratory pressures were measured during a maximal effort for 3 times. The highest value was recorded as cmH2O and also expressed as a percentage of predicted normal values.
Peripheral muscle strength | baseline (pre-operative), 4th and 8th post-operative week
  Knee extension, shoulder flexion and abduction were assessed with a handheld dynamometer. Three maximal isometric contractions are performed. The highest value during the preserved max tension for 1 s was recorded in kg.
Physical performance | baseline (pre-operative), 4th and 8th post-operative week
  30-s Sit-to-Stand Test (STST) provided the number of stands completed with the arms folded across the chest in 30 s. Each functional test was performed twice, in a standardized order, with a 5-min resting period and the best score was recorded.
Functional exercise capacity | baseline (pre-operative), 4th and 8th post-operative week
  Functional exercise capacity was determined by 6-minute walk test (6MWT). The distance covered in 6 minutes along a 30-meters corridor was recorded in meters (6MWD). The predicted 6MWD is calculated using the reference equations.

SECONDARY OUTCOMES:
Fatigue | baseline (pre-operative), 4th and 8th post-operative week
  The 20-item patient-assessed questionnaire Turkish version of Checklist Individual Strength (CIS-T) was used to assess four qualitatively different and relevant aspects of fatigue. Each item is scored on a 7-point Likert scale.
Health-related Quality of Life | baseline (pre-operative), 4th and 8th post-operative week
  HRQoL was measured by Short-Form 36 as a generic tool and The Liver Disease Symptom Index 2.0 as a disease-specific 24-item assessment tool to evaluate the effect of symptoms and their severity on daily activities of patients with chronic liver disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Hospital Groups, Istanbul, Turkey (Türkiye)